CLINICAL TRIAL: NCT04119050
Title: Efficacy and Safety of M281 in Adults With Warm Autoimmune Hemolytic Anemia: A Multicenter, Randomized, Double-blind, Placebo-controlled Study With a Long-term Open-label Extension
Brief Title: Efficacy and Safety of M281 in Adults With Warm Autoimmune Hemolytic Anemia
Acronym: ENERGY
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108987; MOM-M281-006 (Other: Janssen Research & Development, LLC); 2019-000720-17 (EudraCT Number); 2023-505321-14-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2019-09-18; First posted 2019-10-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Warm Autoimmune Hemolytic Anemia
Keywords: Warm Autoimmune Hemolytic Anemia; M281 (Nipocalimab); wAIHA; JNJ-80202135

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- M281 administered every 4 weeks (double-blind period) (Experimental): Participants will receive M281 administered every 4 weeks alternating with placebo every 4 weeks during the 24 weeks double-blind period.
  Interventions: Drug: M281; Drug: Placebo
- M281 administered every 2 weeks (double-blind period) (Experimental): Participants will receive M281 administered every 2 weeks during the 24 weeks double-blind period.
  Interventions: Drug: M281
- Placebo administered every 2 weeks (double-blind period) (Experimental): Participants will receive M281 matching placebo administered every 2 weeks during the 24 weeks double-blind period.
  Interventions: Drug: Placebo
- M281 administered every 4 weeks (open-label extension period) (Experimental): Participants will receive M281 administered every 4 weeks during the 144 weeks open-label extension period.
  Interventions: Drug: M281
- M281 administered every 2 weeks (open-label extension period) (Experimental): Participants will receive M281 administered every 2 weeks during the 144 weeks open-label extension period.
  Interventions: Drug: M281

INTERVENTIONS:
Drug: M281 — M281 injection administered as intravenous infusion
  Other Names: Nipocalimab, JNJ-80202135
  Arms: M281 administered every 2 weeks (double-blind period); M281 administered every 2 weeks (open-label extension period); M281 administered every 4 weeks (double-blind period); M281 administered every 4 weeks (open-label extension period)
Drug: Placebo — Placebo administered as intravenous infusion
  Arms: M281 administered every 4 weeks (double-blind period); Placebo administered every 2 weeks (double-blind period)

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of M281 in participants with warm autoimmune hemolytic anemia (wAIHA).

DETAILED DESCRIPTION:
The study consists of a 24-week double-blind, placebo control period, a 144-week open-label extension period and follow-up period of 8 weeks after last study drug administration. Eligible participants will be randomized to placebo or nipocalimab (2 dose levels) during the double-blind period and nipocalimab (2 dose levels) during the open-label extension period.

ELIGIBILITY:
Inclusion criteria:

* Participants greater than or equal to (>=)18 years of age
* Have been diagnosed with warm autoimmune hemolytic anemia (wAIHA) for at least 3 months, and are currently receiving treatment for wAIHA or have previously received treatment for wAIHA (treatment-naive participants are not eligible)
* Participants must be able to understand and voluntarily provide written informed consent to participate in the study and comply with all study procedures

Exclusion criteria:

* Participants must not be pregnant or breastfeeding
* Participants must not have other clinically relevant abnormalities currently or in their history that the Investigator would deem them ineligible to participate
* Have been diagnosed with cold antibody autoimmune hemolytic anemia (AIHA), cold agglutinin syndrome, mixed type (that is, warm and cold) AIHA, or paroxysmal cold hemoglobinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Durable Response of Improvement in Hemoglobin (Hgb) | Up to Week 20 of the double-blind period

SECONDARY OUTCOMES:
Change From Baseline in the Total Score From the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scale at the Time of Durable Response | Baseline (Day 1, Week 0) through Week 24
  The FACIT-Fatigue is a self-administered 13-item questionnaire that assess patient-reported fatigue associated with chronic illness therapy. It assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from baseline score indicates an improvement.
Change From Baseline in the Total Score From the FACIT-Fatigue Scale at the end of the Double-blind Period (Week 24) | Baseline (Day 1, Week 0) through Week 24 of the double-blind period
  The FACIT-Fatigue is a self-administered 13-item questionnaire that assess patient-reported fatigue associated with chronic illness therapy. It assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from baseline score indicates an improvement.
Change from Baseline in Average Daily Dose of Prednisone or Equivalent | Baseline (Day 1, Week 0) and at Week 24
  Change from baseline in average daily dose of prednisone or equivalent at week 24 among participants on prednisone or equivalent at baseline will be reported.
Number of Participants That Simultaneously Attain Normal Lactate Dehydrogenase, Haptoglobin, and Indirect Bilirubin Levels at a Minimum of 3 Consecutive Visits After Baseline | Baseline (Day 1, Week 0) through Week 24
Percentage of Participants who Experience at Least a 2 g/dL Increase in Hgb From Baseline and Normalization of Lactate Dehydrogenase, Haptoglobin, and Indirect Bilirubin at any Time During the Study | Baseline (Day 1, Week 0) through Week 24
Percentage of Participants who Experience at Least a 2 g/dL Increase in Hgb From Baseline and Normalization of Lactate Dehydrogenase, Haptoglobin, and Indirect Bilirubin at 3 Consecutive Visits | Baseline (Day 1, Week 0) through Week 24
Percentage of Participants who Achieve the Durable Response in Improvement of Hgb During the Double-blind Period and Maintain that Response for Up to 24 Weeks, Without the Need of Rescue Therapy | Up to 24 weeks
  Percentage of participants who achieve the durable response in improvement of Hgb during the double-blind period and maintain that response for up to 24 weeks, without the need of rescue therapy will be reported.
Change From Baseline in Hgb Concentration | Baseline (Day 1, Week 0) through Week 24
Change From Baseline in Reticulocyte Count | Baseline (Day 1, Week 0) through Week 24
Change From Baseline in Hemolytic Marker - Lactate Dehydrogenase | Baseline (Day 1, Week 0) through Week 24
Change From Baseline in Hemolytic Marker - Haptoglobin | Baseline (Day 1, Week 0) through Week 24
Change From Baseline in Hemolytic Marker - Indirect Bilirubin | Baseline (Day 1, Week 0) through Week 24
Time to Hgb Response | Baseline (Day 1, Week 0) through Week 24
Mean Time During Which the Primary Endpoint is Maintained | Baseline (Day 1, Week 0) through Week 24
Change From Baseline in the Total Score, Item Scores, and Impact and Experience Domains From the FACIT-Fatigue Scale | Baseline (Day 1, Week 0) through Week 24 of the double-blind period
  The FACIT-Fatigue scale is a 13-item self-administered questionnaire that assesses both the physical and functional consequences of fatigue. Each question is answered on a 5-point scale, where 0 means "not at all," and 4 means "very much." The FACIT-Fatigue scale score ranges from 0 to 52, with higher scores denoting lower levels of fatigue. A positive change from baseline score indicates an improvement.
Change From Baseline in EuroQol 5-dimension 5-level ( EQ-5D-5L) Scale Score | Baseline (Day 1, Week 0) through Week 24
  The EQ-5D-5L quality of life questionnaire will be used to assess health related quality of life status. The 5 dimensions are mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each dimension is rated by the patient on a 5 level scale (no problems, slight problems, moderate problems, severe problems, extreme problems).
Change From Baseline in Medical Outcomes Study Short Form 36 Item Health Survey Version 2 Acute (SF-36v2) Score | Baseline (Day 1, Week 0) through Week 24
  The SF-36v2 will be used to assess general quality of life. The 36 items on the SF-36 health survey encompass the following 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The 8 domains can be aggregated into 2 summary scales that reflect physical and mental health: a physical component summary (PCS) and a mental component summary (MCS). Responses to all items are rated on a 3-, 5- or 6-point Likert scale. Higher scores indicate a higher level of functioning. A positive change from baseline score indicates an improvement.
Change From Baseline in Patient Global Impression of Severity (PGIS) | Baseline (Day 1, Week 0) through Week 24
  The PGIS will be used to assess the severity of warm autoimmune hemolytic anemia (wAIHA) fatigue symptoms. The PGIS is a 5-point response scale. Participant will be asked to rate their fatigue over the past 7 days using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe.
Patient-reported Status As Assessed by Patient Global Impression of Change (PGIC) Scale Score | At Week 24
  The PGIC will assess if there has been an improvement or decline in patient-reported status since the beginning of the treatment. The PGIC is a 7-point response scale. Participants will be asked to rate their current fatigue as compared to when they started the study, using the following 7-point scale: 1 = Much better, 2 = Moderately better, 3 = A little better, 4 = No change, 5 = A little worse, 6 = Moderately worse, and 7 = Much worse.
Hgb Range at Steady State | Baseline (Day 1, Week 0) through Week 24
  It will be estimated using a model-based longitudinal analysis of Hgb/hemolysis parameters in relationship to IgG level and dose regimen.
Absolute Change from Baseline in Average Daily Dose of Prednisone or Equivalent | Baseline (Day 1, Week 0) and at Week 24
  Absolute change from baseline in average daily dose of prednisone or equivalent at Week 24 among all participants will be reported.
Percentage of participants who Achieve Corticosteroid Reduction to less than or equal to (<=) 7.5 milligrams per day (mg/day) of Oral Prednisone (or Equivalent), Among Participants with Prednisone or Equivalent greater than (>) 7.5 mg/day at Baseline | At Week 24
  Percentage of participants who achieve corticosteroid reduction to <= 7.5 mg/day of oral prednisone (or equivalent) at Week 24 of the double-blind period, among participants with prednisone or equivalent >7.5 mg/day at baseline will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (171):
- United States (29):
  - MemorialCare Medical Group, Fountain Valley, California
  - University of Southern California, Los Angeles, California
  - Compassionate Cancer Care, Riverside, California
  - American Institute of Research, Whittier, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - GNP Research, Cooper City, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - 21st Century Oncology, Jacksonville, Florida
  - Lakes Research, Miami Lakes, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Children's Research Institute, St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Alliance for Multispeciality Research, Merriam, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Henry Ford Medical Center, Detroit, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Montefiore Medical Center, Lake Success, New York
  - Monter Cancer Center, Lake Success, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Taussig Cancer Insititute Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University- James Cancer Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Northwest Medical Specialists, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Brazil (14):
  - Hospital das Clínicas da Faculdade de Medicina de Botucatu, Botucatu
  - Impar Servicos Hospitalares S/A - Hospital Brasilia, Brasília
  - CTO Centro de Tratamento Oncologico Unidade Belem, Campinas
  - Hospital Das Clinicas Da Universidade Federal De Goias, Goiânia
  - Complexo Hospitalar de Niteroi, Niterói
  - Oncoclinicas - Unidade OC Oncoclinicas Multihemo Ilha do Leite, Recife
  - Nucleo de Oncologia da Bahia, Salvador
  - Hospital Sao Rafael, Salvador
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Hospital Santa Marcelina, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- China (16):
  - Beijing Chao-yang Hospital, Capital Medical University, Beijing
  - Peking University People's Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital of Sichuan University, Chengdu
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Hainan General Hospital, Haikou
  - First Affiliated Hospital Medical School of Zhejiang University, Hangzhou
  - Lanzhou University Second Hospital, Lanzhou
  - Jiangsu Province Hospital, Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Shanghai Zhongshan Hospital, Shanghai
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University General Hospital, Tianjin
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Ustav Hematologie A Krevni Transfuze, Prague
- Egypt (6):
  - Mansoura University Hospital, Al Mansurah
  - Alexandria University Hospital, Alexandria
  - Cairo university, Cairo
  - Ain Shams University Hospital, Cairo
  - National Cancer Institute, Cairo
  - Nasser institute Hospital, Cairo
- France (6):
  - ICH Hopital A. Morvan, Brest
  - CHU Dijon Bourgogne, Dijon
  - CHU Grenoble, La Tronche
  - CHU Nantes - Hotel Dieu, Nantes
  - CHU De Poitiers, Poitiers
  - CHRU Hopital Sud, Rennes
- Germany (3):
  - Onkologische Schwerpunktpraxis, Berlin
  - Universitatsklinikum Essen, Essen
  - Rotkreuzklinikum München, München
- Greece (6):
  - General Hospital of Athens G Gennimatas, Athens
  - Laiko General Hospital of Athens, Athens
  - Attikon University General Hospital of Attica, Athens
  - University Hospital Of Larissa, Larissa
  - University General Hospital of Rio Patras, Pátrai
  - University General Hospital of Thessaloniki, Thessaloniki
- Hungary (5):
  - Semmelweis Egyetem, Budapest
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Gyõr
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
- Israel (8):
  - Ha'Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Hospital Sanz Medical Center Laniado Hospital, Kiryat Tzanz
  - Rabin Medical Center, Beilinson Hospital, Petach Tikvah
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - PO C e G Mazzoni AST Ascoli Piceno, Ascoli Piceno
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione Garibaldi, Catania
  - AOU Policlinico G Rodolico S Marco, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara, Novara
  - Umberto I Policlinico di Roma, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
  - Azienda Ulss 8 Berica- Ospedale Di Vicenza, Vicenza
- Japan (12):
  - Fukushima Medical University Hospital, Fukushima
  - Saitama Medical University Hospital, Iruma-gun
  - St Marianna University Hospital, Kanagawa
  - Japan Community Health care Organization Kyushu Hospital, Kitakyusyu-Shi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Ogaki Municipal Hospital, Ōgaki
  - Sapporo Medical University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Osaka University Hospital, Suita
  - Toyama Prefectural Central Hospital, Toyama
  - Wakayama Medical University Hospital, Wakayama
  - Tottori University Hospital, Yonago
- Malaysia (7):
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah, Johor Bharu
  - Hospital Queen Elizabeth, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Sunway Medical Centre, Petaling Jaya
- Netherlands (3):
  - Amsterdam Universitair Medische Centra Locatie Vrije Universiteit Medisch Centrum, Amsterdam
  - Academic Medical Centre Amsterdam, Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
- Poland (6):
  - Interhem, Bialystok
  - Klinika Hematologii i Transplantologii, UCK, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Szpital Wojewodzki w Opolu, Opole
  - MTZ Clinical Research Powered by Pratia, Warsaw
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (20):
  - Hosp. Univ. Principe de Asturias, Alcalá de Henares
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Complejo Asistencial Univ. de Burgos, Burgos
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Virgen Del Rocio, Málaga
  - Hosp. Son Llatzer, Palma de Mallorca
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Univ. Miguel Servet, Zaragoza
- Ukraine (5):
  - Cherkassy Regional Oncology Dispensary, Department of Hematology, Cherkassy
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk City Multifield Clinical Hospital # 4, Dnipro
  - Medical Center 'Ok Clinic' of LLC 'International Institute of Clinical Studies', Kyiv
  - Kyiv City Clinical Hospital #9, Department of infectious diseases, Kyiv
  - Ternopil University Hospital of Ternopil Regional Council, Ternopil
- United Kingdom (6):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu AP, Cheuk DK. Disease-modifying treatments for primary autoimmune haemolytic anaemia. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012493. doi: 10.1002/14651858.CD012493.pub2. PMID 33786812
- See also: Participant recruitment poster — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108987&attachmentIdentifier=8895a4ed-7f9f-4d12-b738-91162ef80bd5&fileName=Energy_Study_Patient_Poster__(1).pdf&versionIdentifier=